CLINICAL TRIAL: NCT01999322
Title: A 6-week Randomised, Double-blind, Parallel-group Trial Evaluating Compatibility and Safety of FIAsp and Insulin Aspart With an External Continuous Subcutaneous Insulin Infusion System in Adult Subjects With Type 1 Diabetes
Brief Title: A Trial Evaluating Compatibility and Safety of FIAsp and Insulin Aspart With an External Continuous Subcutaneous Insulin Infusion System in Adult Subjects With Type 1 Diabetes
Acronym: onset® 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3931; 2013-002233-37 (EudraCT Number); U1111-1143-2316 (Other: WHO)
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Results first posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FIAsp (Experimental): The trial duration is approximately 13 weeks and consists of a 1-week screening period, a 2-week run-in period, a 6-week treatment period and 1 week plus a 30-day follow-up period
  Interventions: Drug: Faster-acting insulin aspart
- Insulin Aspart (Active Comparator): The trial duration is approximately 13 weeks and consists of a 1-week screening period, a 2-week run-in period, a 6-week treatment period and 1 week plus a 30-day follow-up period
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Administered subcutaneously (s.c., under the skin). Dose individually adjusted.
  Arms: FIAsp
Drug: insulin aspart — Administered subcutaneously (s.c., under the skin). Dose individually adjusted.
  Arms: Insulin Aspart

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The aim of this trial is to evaluate compatibility and safety of FIAsp (faster-acting insulin aspart) and insulin aspart (NovoRapid®) with an external continuous subcutaneous insulin infusion (CSII) system in adult subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age at least 18 years at the time of signing inform consent
* Type 1 diabetes mellitus (diagnosed clinically) for at least 12 months at the time of screening (Visit 1)
* Currently treated with insulin aspart, insulin lispro or insulin gluisine for at least 3 months prior to screening (Visit 1)
* Using an external CSII system for the previous 6 months prior to screening (Visit 1)
* HbA1c (glycosylated haemoglobin) below or equal to 9.0% as assessed by central laboratory
* Body Mass Index (BMI) 20.0-35.0 kg/m^2

Exclusion Criteria:

* History of diabetic ketoacidosis (DKA) episodes requiring hospitalization within 6 months prior to screening (Visit 1)
* History of abscess at the infusion site within 6 months prior to screening (Visit 1)
* Hypoglycaemic unawareness as judged by the Investigator or history of severe hypoglycaemic episodes requiring hospitalization within the last 6 months prior to screening (Visit 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-11-19 (Actual); Primary Completion 2014-05-14 (Actual); Study Completion 2014-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Novo Nordisk Investigational Site, Atlanta, Georgia, United States
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Background] Zijlstra E, Demissie M, Graungaard T, Heise T, Nosek L, Bode B. Investigation of Pump Compatibility of Fast-Acting Insulin Aspart in Subjects With Type 1 Diabetes. J Diabetes Sci Technol. 2018 Jan;12(1):145-151. doi: 10.1177/1932296817730375. Epub 2017 Sep 18. PMID 28918652
- [Result] Eric Zijlstra, Marek Demissie et al. Compatibility and Safety of Faster-Acting Insulin Aspart used in Continuous Subcutaneous Insulin Infusion Therapy in Patients with Type 1 Diabetes. ENDO-2016-98th Annual Meeting of the Endocrine Society 3 June 2016 http://press.endocrine.org/doi/abs/10.1210.endo-meetings.2016.DGM.22.FRI-697
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at two sites in two countries as follows: USA: one site; Germany: one site.
Pre-assignment Details: Eligible subjects previously treated with a rapid acting insulin analogue were to stay on their own NovoRapid®, insulin lispro or insulin glulisine in the screening period after which the all subjects received NovoRapid®, with no additional antidiabetics allowed, for a 2-week run-in period prior to randomisation.
Groups:
- Faster-acting Insulin Aspart: Subjects received faster-acting insulin aspart for a duration of 6 weeks. Faster-acting insulin aspart was provided in 100U/ml 3 mL Penfill® and administered in accordance with the instructions provided by the pump manufacturer, preferably in the abdomen, by subcutaneous infusion. The insulin dose adjustments were made based on frequent glucose measurements during contacts with the investigator. The following glycaemic targets were recommended: preprandial and bedtime glucose: below 6.0 mmol/L (108 mg/dL) and 2-hr postprandial glucose: below 7.8 mmol/L (140 mg/dL). A 2:1 randomisation following the screening period was selected in order to ensure adequate exposure to faster-acting insulin aspart.
- NovoRapid®: Subjects received NovoRapid® for a duration of 6 weeks. NovoRapid® was provided in 100U/ml 3 ml Penfill® and administered in accordance with the instructions provided by the pump manufacturer, preferably in the abdomen, by subcutaneous infusion. The insulin dose adjustments were made based on frequent glucose measurements during contacts with the investigator. The following glycaemic targets were recommended: preprandial and bedtime glucose: below 6.0 mmol/L (108 mg/dL) and 2 hr postprandial glucose: below 7.8 mmol/L (140 mg/dL).
Period: Overall Study
Arm/Group | Faster-acting Insulin Aspart | NovoRapid®
Started | 25 | 12
Completed | 24 | 12
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: included all randomised subjects. In exceptional cases subjects could be excluded from the full analysis set. In such cases the reason for exclusion was to be justified and documented. Safety analysis set: includes all subjects receiving at least one dose of the investigational product or its comparator.
Groups:
- Total: Total of all reporting groups
Arm/Group | Faster-acting Insulin Aspart | NovoRapid® | Total
Number analyzed (Participants) | 25 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (14.6) | 34.7 (9.1) | 44.3 (14.6)
Age, Customized [Number; unit: participants]
  18-64 | 19 | 12 | 31
  65-84 | 6 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 14 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Microscopically Confirmed Episodes of Infusion Set Occlusions
Description: The number of microscopically confirmed episodes of infusion set occlusions during 6 weeks of treatment. Episodes of infusion set occlusions were confirmed by microscopic examination of the infusion sets at each routine weekly visit and infusion sets that had been changed prematurely because of leakage, unexplained hyperglycaemia or suspicion of occlusion (observation of a plug).
Time Frame: During 6 weeks of treatment
Population: FAS: included all randomised subjects. In exceptional cases subjects could be excluded from the full analysis set. In such cases the reason for exclusion was to be justified and documented. Subjects in the full analysis set contribute to the evaluation "as randomised".
Measure: Number; unit: Episodes
Arm/Group | Faster-acting Insulin Aspart | NovoRapid®
Number analyzed (Participants) | 25 | 12
Episodes | 0 | 0

2. Secondary Outcome: Number of Unexplained Episodes of Hyperglycaemia (Confirmed by Self-measured Plasma Glucose (SMPG))
Description: Unexplained hyperglycaemia was defined as a confirmed plasma glucose value ≥ 16.7 mmol/L (300 mg/dL) and was unexplained (i.e., no apparent medical, dietary, insulin dosage or pump failure reason)
Time Frame: During 6 weeks of treatment
Measure: Number; unit: events
Arm/Group | Faster-acting Insulin Aspart | NovoRapid®
Number analyzed (Participants) | 25 | 12
events | 28 | 16

3. Secondary Outcome: Number of Episodes of Possible Infusion Set Occlusions
Description: Episodes of possible infusion set occlusions were defined as infusion sets changed due to suspicion of occlusion, leakage or unexplained hyperglycaemic episode. Possible occlusion excluded technical reasons. This endpoint was calculated from the recorded date/times of changes of infusion set combined with the subjects' own assessment.
Time Frame: During 6 weeks of treatment
Measure: Number; unit: Episodes
Arm/Group | Faster-acting Insulin Aspart | NovoRapid®
Number analyzed (Participants) | 25 | 12
Episodes | 7 | 0

4. Secondary Outcome: Number of Premature Infusion Set Changes
Description: A premature infusion set change was defined as not being a routine change. This was defined as an infusion set changed at home due to "suspicion of occlusion", "leakage", "unexplained hyperglycaemic episode", "infusion site reaction", "technical reason", or "other". The change of infusion set at a site visit was considered a routine change unless an occlusion was actually suspected at the site.
Time Frame: During 6 weeks of treatment
Measure: Number; unit: Episodes
Arm/Group | Faster-acting Insulin Aspart | NovoRapid®
Number analyzed (Participants) | 25 | 12
Episodes | 21 | 4

ADVERSE EVENTS:
Time Frame: A treatment emergent adverse event is defined as en event that has onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment.
Description: Safety Analysis Set: includes all subjects receiving at least one dose of the investigational product or its comparator.
Arm/Group | Faster-acting Insulin Aspart | NovoRapid®
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/12
Other Adverse Events (participants affected / at risk) | 9/25 | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faster-acting Insulin Aspart (N=25) | NovoRapid® (N=12)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was designed in accordance with the draft FDA guideline dated 1985, that 15-20 subjects with diabetes given the modified insulin should be included for 6 weeks. However the trial was not powered to detect differences between treatments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property"